CLINICAL TRIAL: NCT01486849
Title: A Phase II, Multicenter, Double-Blind, Randomized, Placebo-Controlled Dose Titration Study to Evaluate the Safety, Tolerability and Pharmacodynamic Effects of CK-2017357 in Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Dose Titration Study to Test Safety and Effects of CK-2017357 in Patients With Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CY 4025
Record Dates: First submitted 2011-11-23; First posted 2011-12-07 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-04

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — CK-2017357; Riluzole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose Titration of CK-2017357 (Group 1) (Experimental): Dose titration of active drug as add-on therapy to riluzole
  Interventions: Drug: CK-2017357; Drug: Riluzole 50 MG
- Matching Placebo (Group 2) (Placebo Comparator): Placebo as add-on therapy to riluzole
  Interventions: Drug: Placebo; Drug: Riluzole 50 MG

INTERVENTIONS:
Drug: CK-2017357 — Total daily oral dose of 250 mg (125 mg BID) of CK-2017357 for 7 days followed by total daily oral dose of 375 mg (125 mg AM and 250 mg PM) for 7 days followed by total daily oral dose of 500 mg (250 mg BID) of CK-2017357 for 7 days
  Other Names: tirasemtiv
  Arms: Dose Titration of CK-2017357 (Group 1)
Drug: Placebo — Matching placebo tablets BID for 21 days
  Arms: Matching Placebo (Group 2)
Drug: Riluzole 50 MG

SUMMARY:
A Phase II, double-blind, randomized, placebo-controlled ascending dose titration study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamic effects of multiple ascending doses of CK-2017357 to an individual patient maximum tolerated dose (MTD), using a within-patient twice daily (BID) dose-titration regimen in ALS patients on 50 mg riluzole once daily (QD).

DETAILED DESCRIPTION:
Patients will be randomized to one of two dosing groups, active CK-2017357 or placebo, in a 3:1 ratio. Prior to study drug dosing, patients will be required to decrease their riluzole dose to 50 mg QD for 7 days; after this 7 day period patients will either receive placebo or start the titration on active CK-2017357 while continuing to take riluzole at 50 mg QD.

Potential patients will be screened to assess their eligibility to enter the study within 21 days prior to Day -7, when they will begin taking riluzole at the decreased dose of 50 mg QD. Patients will be randomized in a 3:1 ratio to CK-2017357 (Group 1) or placebo (Group 2). On Day 1, patients will begin taking a total daily dose of 250 mg (125 mg BID) of CK-2017357 or matching placebo tablets BID for 7 days. Then they will take a total daily dose of 375 mg (125 mg morning [AM] and 250 mg evening [PM]) of CK-2017357 or matching placebo tablets BID for 7 days, and finally, they will take a total daily dose of 500 mg (250 mg BID) of CK-2017357 or matching placebo tablets BID for 7 days. A final dose of 250 mg of CK-2017357 or placebo will be taken in the morning on Day 22 at the study site.

Dose-escalation of CK-2017357 or placebo may be stopped, or the dose reduced to a lower level, based on tolerability. All patients who return to a lower dose will stay on that dose for the remainder of the study.

Patients will remain on the decreased dose of riluzole until the follow-up visit approximately 7 days after Day 22.

ELIGIBILITY:
Inclusion Criteria:

1. Able to comprehend and willing to sign an Informed Consent Form (ICF)
2. Males or females 18 years of age or older
3. A diagnosis of familial or sporadic ALS (defined as meeting the possible, laboratory-supported probable, probable, or definite criteria for a diagnosis of ALS according to the World Federation of Neurology El Escorial criteria)
4. Maximum voluntary grip strength in at least one hand between 10 & 40 pounds (females) and 10 & 60 pounds (males)
5. Able to swallow tablets with water
6. Currently taking and tolerating a stable dose of 50 mg BID riluzole
7. Willing and able to reduce daily dose of riluzole to 50mg QD for 5 weeks
8. Not currently taking or willing and able to remain off theophylline-containing medications during study participation
9. Patient has a caregiver who is capable of observing and reporting patient status
10. Upright Slow Vital Capacity (SVC) >50% of predicted for age, height, and sex
11. Able to perform pulmonary function tests

Exclusion Criteria:

1. Life expectancy <3 months
2. Receipt of investigational study drug within 30 days or 5 half-lives of the prior agent, whichever is greater, prior to dosing
3. Any prior treatment with CK-2017357
4. Any use of non-invasive positive pressure ventilation (NIPPV), such as Continuous Positive Airway Pressure (CPAP) or Bilevel Positive Airway Pressure (BiPAP)

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | approximately 29 days

SECONDARY OUTCOMES:
Change from baseline in score on the Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) | 22 days
  An instrument for evaluating the functional status of patients with ALS. Minimum score is 0 and maximum score is 40. The higher the score the more function is retained. This will be administered at Screening, Day -7, Day 1, Day 15 and Day 22.
Change from baseline in scores on tests of maximum handgrip strength and handgrip fatigue | 22 days
  Measured using the DynEx Electronic Hand Dynamometer. Patients asked to squeeze the device with the maximum possible force to establish the maximum voluntary contraction. Handgrip fatigue is then measured. Patient is asked to squeeze the device until they can no longer stay above 60% of target or 120 seconds. This will be measured at Screening, Day -7, Day 1, Day 15 and Day 22.
Change from baseline in scores on tests of muscle strength | 22 days
  Muscle strength is measured using Hand Held Dynamometry. A series of assessments are done on different muscle groups. This will be measured at Day -7, Day 1, and Day 22.
Change from baseline in scores on tests of Timed Up and Go | 22 days
  TUG is measured by timing how long it takes for a subject to stand up from a chair, walk 10 feet, turn around, walk back to the chair and sit down. This will be measured at Day -7, Day 1, and Day 22.
Change from baseline in scores on tests of Sniff Nasal Inspiratory Pressure (SNIP) | 22 days
  SNIP will be measured using the Micro Medical Respiratory Pressure Meter (MicroRPM) at Screening, Day -7, Day 1, Day 15 and Day 22.
Change from baseline in scores on tests of Slow Vital Capacity (SVC) | 22 days
  SVC will be measured using the ndd EasyOne Spirometer System at Screening, Day -7, Day 1, Day 15 and Day 22.
Change from baseline in scores on tests of Maximum Voluntary Ventilation (MVV) | 21 days
  MVV will be measured using the EasyOne Spirometer System at Screening, Day -7, Day 1, Day 15 and Day 22.
Change from baseline in Patient Global Assessment | 22 days
  Patients will be asked to assess whether they feel the same, better or worse as compared to how they felt at pre-dose on Day 1
Change from baseline in Investigator Global Assessment | 22 days
  Investigator will assess whether the patient appears the same, better or worse as compared to the patient's status at pre-dose on Day 1.
Evaluate the pharmacokinetics of CK-2017357 | Day 1, Day 15, and Day 22
  Plasma levels of CK-2017357 will be measured at pre-dose, and at 2 and 4 hours post AM dose
Evaluate the pharmacokinetics of riluzole in patients receiving CK-2017357 | Day 1, Day 15, and Day 22
  Plasma levels of riluzole will be measured at pre-dose and at 2 and 4 hours post AM dose

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Shefner, MD, PhD, Study Chair — State University of New York - Upstate Medical University
Locations (11):
- United States (11):
  - University of California at San Francisco, Fresno Campus, Central California Neurological Institute, Fresno, California
  - Coordinated Clinical Research, La Jolla, California
  - University of California at Irvine, ALS and Neuromuscular Center, Orange, California
  - Hospital for Special Care, New Britain, Connecticut
  - Massachusetts General Hospital, Neurology Clinical Trials Unit, Charlestown, Massachusetts
  - Washington University, St Louis, Missouri
  - Cornell Faculty, Hospital for Special Surgery, New York, New York
  - Duke University School of Medicine, Division of Neurology, Durham, North Carolina
  - Ohio State University, Department of Neurology, Columbus, Ohio
  - Providence ALS Center, Portland, Oregon
  - University of Texas Health Science Center, Department of Neurology, San Antonio, Texas